CLINICAL TRIAL: NCT03375294
Title: Exploring Nitrous Oxide Effects for Post Traumatic Stress Disorder (PTSD)
Acronym: tN2O
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41822
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nitrous Oxide (Experimental): PTSD patients in this arm will receive a single inhalation dose of 50% nitrous oxide and 50% oxygen for 1 hour
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — One hour inhalation of 50% nitrous oxide, an odorless, colorless gas FDA approved as an induction agent for dental sedation

SUMMARY:
The purpose of this study is to understand nitrous oxide effects in post traumatic stress disorder (PTSD)

DETAILED DESCRIPTION:
Post traumatic stress disorder (PTSD) is a disabling mental health disorder that impacts the lives of individuals. This study aims to understand nitrous oxide's effects in PTSD.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* Veterans of the United States Uniformed Services
* primary diagnosis of PTSD
* sufficient severity of PTSD symptoms
* fluency in English
* capacity to provide informed consent

Exclusion Criteria:

* psychiatric or medical conditions that make participation unsafe
* pregnant or nursing females
* allergy to nitrous oxide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Veterans Affairs Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varias A, van Roessel P, Parsiani M, Filippou-Frye M, Neylan TC, Nagele P, Yesavage J, Clark JD, Rodriguez CI. Does Nitrous Oxide Help Veterans With Posttraumatic Stress Disorder? A Case Series. J Clin Psychiatry. 2020 Jun 30;81(4):20l13393. doi: 10.4088/JCP.20l13393. No abstract available. PMID 32609959
- See also: Rodriguez Lab Website — http://rodriguezlab.stanford.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrous Oxide
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: Patients given CAPS-5 (Clinician Administered PTSD Scale for DSM-5), a 30-item structured interview that can be used to assess PTSD symptoms over the past week. For the CAPS-5 the minimum units are 0 and maximum units on the total scale are 80. The higher the number on the CAPS-5, the more severe the symptoms. Response was defined as at least a 12 point reduction on the CAPS-5
Time Frame: Baseline and 1 week post inhalation
Population: 3 Veteran outpatients ages 31, 43, and 46 who met PTSD criteria of at least moderate symptoms severity (CAPS-5 score equal or greater than 40)
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 week
Description: Does not differ.
Arm/Group | Nitrous Oxide
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide (N=3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Poor concentration (Nervous system disorders) | 2 (2)
Decreased energy (Gastrointestinal disorders) | 1 (1)
General malaise (Nervous system disorders) | 1 (1)
Fingers tingling (Nervous system disorders) | 1 (1)
Body warmth (Nervous system disorders) | 1 (1)
Increased perspiration (Nervous system disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Restlessness (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03375294/Prot_SAP_000.pdf